CLINICAL TRIAL: NCT05928221
Title: Clinical Safety, Feasibility, and Economic Viability of Performing Percutaneous Deep Vein Thrombectomy With the QuickClear Thrombectomy System in an Office Interventional Suite for Acute Lower Extremity Deep Vein Thrombosis (DVT)
Brief Title: Post Market Registry Study of the Philips QuickClear Mechanical Thrombectomy System
Status: Active, not recruiting | Type: Observational
Sponsor: Paul J. Gagne (Other)
Responsible Party: Sponsor-Investigator, Paul J. Gagne, President, Vascular Breakthroughs, LLC, Vascular Care CT, PLLC
Organization: Vascular Care CT, PLLC (Other)
Other Study IDs: CP-001
Record Dates: First submitted 2023-06-12; First posted 2023-07-03 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Acute Deep Venous Thrombosis of Ileofemoral Vein
MeSH Terms: interventions — Thrombectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Thrombectomy — removal of fresh soft emboli and thrombi from the vessels of the venous system
  Other Names: QuickClear Mechanical Thrombectomy system

SUMMARY:
A post-market study of the QuickClear Mechanical Thrombectomy system used for the removal of acute Deep Vein Thrombosis (DVT) from the deep veins of legs in the setting of an office interventional suite.

DETAILED DESCRIPTION:
The QuickClear Mechanical Thrombectomy system will be used in accordance with the Instruction for Use (IFU) to remove acute, symptomatic occlusive common femoral, external iliac or common iliac DVT or occlusive above and below knee popliteal DVT in an office based interventional suite. The intent of this post-market observational study is to further assess long-term safety and effectiveness of patients treated with the QuickClear Mechanical Thrombectomy system and to assess the feasibility of performing deep vein thrombectomy procedures in the office interventional suite.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Non-Pregnant Female, age 18 to 89.
2. For females of reproductive potential: negative pregnancy test ≤ 7 days before the procedure, use of highly effective contraception (abstinence is acceptable) for 12 months after the study treatment.
3. Onset of acute DVT symptoms of 14 days or less in the target limb.
4. Ability to take oral medication and be willing to adhere to the prescribed anti- coagulant regiment.
5. Occlusive DVT (confirmed by either venous duplex ultrasound or CT venogram) spanning at least one of the following:

   1. the iliac and/or common femoral vein. Extension into the femoral vein and/or profunda vein is allowed. OR
   2. the entire popliteal vein (above and below knee). Extension into the femoral vein and/or tibial veins is allowed.
6. People who have scheduled or will be scheduled for treatment with the QuickClear Mechanical Thrombectomy system
7. Symptomatic DVT defined as meeting at least one of the following clinical indicators:

   1. rVCSS Pain Score ≥2
   2. New edema of calf or thigh (CEAP ≥3)

Exclusion Criteria:

1. Non-ambulatory status prior to DVT occurrence.
2. Inability to lie in supine or prone under local anesthesia with moderate sedation for procedure.
3. In the contralateral (non-study) leg: symptomatic DVT that, in the operating physician's opinion, will require treatment in the following 30 days.
4. Critical limb ischemia with ulcer, gangrene, or rest pain (i.e., above symptoms or findings and ankle-brachial index <0.5, absolute ankle pressure <50 mm Hg or absolute toe pressure <30 mmHg).
5. Pulmonary embolism (PE) defined as either massive (systolic blood pressure < 90 mm Hg and/or patient on IV vasoactive medication to support blood pressure), or intermediate high-risk PE, as defined by the European Society Guideline on management of PE. Low-risk PE and/or intermediate low-risk PE can be enrolled.
6. Inability to tolerate contemporary venous intervention procedure due to severe dyspnea or acute systemic illness.
7. Allergy, hypersensitivity, or thrombocytopenia from heparin, iodinated contrast, except for mild-moderate contrast allergies for which steroid pre-medication can be used.
8. History of, or active heparin-induced thrombocytopenia (HIT).
9. Hemoglobin ≤9.0 mg/dl, INR>1.6 before starting anticoagulation, or platelets < 100,000/ml. Moderate renal impairment in diabetic patients (eGFR <60 ml/min) or severe renal impairment in non-diabetic patients (eGFR< 30 ml/min).
10. Active bleeding, recent (< 3 mo) GI bleeding, severe liver dysfunction, bleeding diathesis.
11. Recent (< 3 mo) internal eye surgery or hemorrhagic retinopathy; recent (<10 days) major surgery, cataract surgery, trauma, cardiopulmonary resuscitation, or other invasive procedure; or obstetrical delivery < 72 hours prior to procedure.
12. History of hemorrhagic stroke or intracranial/intraspinal bleed, tumor, vascular malformation, aneurysm.
13. Active cancer with a life expectancy of < 1 year.
14. Severe hypertension on repeated readings (systolic blood pressure > 180 mm Hg or diastolic blood pressure >105 mmHg). This can be treated, and blood pressure must be stable before venous access is obtained (systolic blood pressure < 150 mmHg, diastolic blood pressure < 100 mm Hg).
15. Pregnant or breastfeeding or plans to become pregnant in the next 12 months.
16. Thrombus of the inferior vena cava (IVC) extending at least one centimeter above the common iliac vein confluence.
17. Inability to obtain venous access.
18. Contraindication to Enoxaparin (e.g., Severe chronic kidney injury, allergic reaction, HIT)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who receive treatment with Philips QuickClear Mechanical Thrombectomy system in accordance with the current approved FDA indication for use as stated in the Instructions for Use (IFU) for acute lower extremity DVT.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-06-14 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Primary Device Effectiveness | Immediately after procedure
  Extent of acute DVT removal overall and in each segment (Common Iliac Vein (CIV), External Iliac Vein (EIV), Common Femoral Vein (CFV), Profunda Femoris Vein (PFV), Femoral Vein (FV), Popliteal (POP) as measured by IVUS and Venography
Change in revised Venous Clinical Severity Score (rVCSS) | 30 days post index procedure
  Improvement of target leg revised Venous Clinical Severity Score (rVCSS)
  Scores range from 0= no disease to 30= severe disease. Change in the rVCSS score is calculated as the follow-up score minus the Baseline score
  . A negative change is associated with improved outcome
Change in Villalta Score | 30 Days Post Index Procedure
  Improvement of the Villalta Score.
  Villalta scores categorize the severity of post-thrombotic syndrome (PTS). Higher score indicates increasing severity of PTS. A score of greater or equal to 5 indicates PTS. PTS severity: total score of 5 to 9, mild PTS; score of 10 to 14, moderate PTS; and score of greater or equal to 15 or venous ulcer present, sever PTS.
  A negative change is associated with improved outcome.
Change in EuroQol-5 Dimension (EQ-5D) Score | 30 Days Post Index Procedure
  Higher score indicates a better quality of life. The questionnaire contains five dimensions where scores rank from 1 (best) to 5 (worst) plus a visual analog scale (VAS) (0=worst health; 100= best health).
  A positive change is associated with improved outcome. Change in EQ-5D scores are calculated as the Follow-up minus the Baseline score.
Primary Safety Endpoint | 12 months post index procedure
  Serious adverse event related to the device, study procedure or secondary procedure to maintain or re-establish patency

SECONDARY OUTCOMES:
Total blood loss during procedure | immediately after index procedure
  The total blood loss for the duration of the procedure will be determined by the volume of blood in the collection bag, measured in milliliters, at the end of the procedure.
Age of Deep Vein occlusive disease | immediately after the procedure
  The Deep Vein occlusive disease will be categorized as one of the following depending on the age of the disease visualized during the procedure: Acute DVT, Acute DVT on chronic scar, chronic scar
Health Economics | 3 months post index procedure
  Analysis of procedural reimbursement versus procedural cost of treatment
Primary patency | 12 months post index procedure
  Primary patency through 12 months of vein segments that were patent (>50% lumen) at end of index procedure
Assisted primary patency | 12 months post index procedure
  required reintervention to maintain patency
Change in revised Venous Clinical Severity Score (rVCSS) | 12 months post index procedure
  Improvement of target leg rVCSS
  Scores range from 0= no disease to 30= severe disease. Change in the rVCSS score is calculated as the follow-up score minus the Baseline score
  . A negative change is associated with improved outcome
Overall patient safety | 12 months post procedure
  Adverse event tracking
Change in Villalta Score | 12 months post index procedure
  Improvement of the Villalta Score.
  Villalta scores categorize the severity of post-thrombotic syndrome (PTS). Higher score indicates increasing severity of PTS. A score of greater or equal to 5 indicates PTS. PTS severity: total score of 5 to 9, mild PTS; score of 10 to 14, moderate PTS; and score of greater or equal to 15 or venous ulcer present, sever PTS.
  A negative change is associated with improved outcome.
Change in EuroQol-5 Dimension (EQ-5D) Score | 12 months post index procedure
  Higher score indicates a better quality of life. The questionnaire contains five dimensions where scores rank from 1 (best) to 5 (worst) plus a visual analog scale (VAS) (0=worst health; 100= best health).
  A positive change is associated with improved outcome. Change in EQ-5D scores are calculated as the Follow-up minus the Baseline score.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Vascular Care Connecticut, Darien, Connecticut
  - The Vascular Care Group, Hyannis, Massachusetts
  - The Vascular Care Group, Leominster, Massachusetts
  - The Vascular Care Group, Plymouth, Massachusetts
  - The Vascular Care Group, Wellesley, Massachusetts
  - The Vascular Care Group, Worcester, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided